CLINICAL TRIAL: NCT04931511
Title: Comparison Between Subacromial Ultrasound Guided and Systemic Steroid Injection for Frozen Shoulder: a Randomized Double Blind Study
Brief Title: Comparison Between Subacromial Ultrasound Guided and Systemic Steroid Injection for Frozen Shoulder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Since the COVID-19 pendemic, the regular follow-up of participant became very hard. The participant were not willing to go back to the hospital for repeat measurement. So we stop the study and plan to redesign the protocol.
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, huang pintong, Director of the department of ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Study 2020-1064
Record Dates: First submitted 2021-04-08; First posted 2021-06-18 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Frozen Shoulder; Shoulder Pain; Bursitis
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Adrenal Cortex Hormones; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluteal muscle injection plus physical therapy group (Experimental): Gluteal muscle injection (corticosteroid 1ml+normal saline 4ml) + Subacromial Ultrasound Guided injection (sodium chloride 5ml) + Physical therapy
  Interventions: Drug: Compound betamethasone Injection(Gluteal muscle injection); Behavioral: Physical therapy
- Subacromial Ultrasound Guided injection plus physical therapy group (Experimental): Gluteal muscle injection(sodium chloride 5ml)) + Subacromial Ultrasound Guided injection(corticosteroid 1ml+normal saline 4ml) + Physical therapy
  Interventions: Drug: Compound betamethasone Injection(Subacromial Ultrasound Guided injection); Behavioral: Physical therapy

INTERVENTIONS:
Drug: Compound betamethasone Injection(Gluteal muscle injection) — Gluteal muscle injection(Compound betamethasone 1ml + Sodium Chloride Injection 4ml) + Subacromial Ultrasound Guided injection(Sodium Chloride Injection 5ml)
  Other Names: corticosteroid
  Arms: Gluteal muscle injection plus physical therapy group
Drug: Compound betamethasone Injection(Subacromial Ultrasound Guided injection) — Gluteal muscle injection (Sodium Chloride Injection 5ml)+ Subacromial Ultrasound Guided injection (corticosteroid 1ml+Sodium Chloride Injection 4ml)
  Other Names: corticosteroid
  Arms: Subacromial Ultrasound Guided injection plus physical therapy group
Behavioral: Physical therapy — paticipant will be teached by the Physicaltherapist to reduce the shoulder pain at home

SUMMARY:
This study aim to compare the efficacy of guteal muscle injection and subacromial ultrasound guided injection to treat frozen shoulder. Firstly, in order to calculate the sample size correctly, we start the preliminary study. Besides, in order to propose clinical new technology which combines the advantages of the two therapies, improve the efficacy ratio of frozen shoulder therapy, and provide a frozen shoulder treatment plan according to health economics.

DETAILED DESCRIPTION:
In recent years, there have been studies suggesting that small doses of corticosteroid systemic medication and joint local injection to treat shoulder sleeve disease is equivalent, frozen shoulder is clinically in addition to shoulder sleeve disease another common cause of shoulder pain disease, local injection of small dose of corticosteroid is a clinically commonly used treatment of frozen shoulder mature therapy, however, because of the risk of joint infection and other serious complications, and it's personnel experience depended and high qualification requirements, resulting in higher treatment costs. However, it has not been widely used in clinical applications and is generally used as a second-line therapy for the treatment of frozen shoulders. There are studies suggesting that joint cavity hormone injection may be mainly effective through its systemic effect, however, there is currently no random blind control study comparing small doses of hormone systemic injection with local injection of shoulder joints to freeze shoulder, if the equivalence of the two can be confirmed through such studies will greatly change the clinical treatment of frozen shoulders, with hip injection and other systemic medication will provide great health economic advantages, and can avoid the inherent risk of joint cavity injection, reduce the social cost of frozen shoulder treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary frozen shoulder
* 2. Older than 18 years of age and less than 75 years of age
* 3. The SHOULDER PAIN VAS SCORE IS GREATER THAN 3 POINTS AND LASTS AT LEAST 1 MONTH AND LESS THAN 9 MONTHS
* 4. The passive activity of the side shoulder joint in at least 2 directions in the three directions of front, internal and outer rotation decreased by more than 30 degrees compared to the side shoulder joint or the normal reference value
* 5. corticosteroid injections were not given within 3 months of visit

Exclusion Criteria:

* 1. A history of trauma, osteoarthritis, tumors, etc.
* 2. Combined shoulder sleeve injury with magnetic resonance or B-mode ultrasound confirmed
* 3. There is a history of corticosteroid injections within 3 months of visit
* 4. Suffer from a partial infection of the side shoulder or other cases where there is a contraindication of shoulder injection
* 5. Both side shoulder joints become ill at the same time
* 6. The patient has not signed an informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The Change of Shoulder Pain and Disability Index (SPADI) | 0,1,2,4,8,12 weeks
  The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

SECONDARY OUTCOMES:
The Change of Numeric Rating Scale for Pain (NRS) (Score: 0-10) | 0,1,2,4,8,12 weeks
  The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. The common format is a horizontal bar or line. Similar to the pain VAS, the NRS is anchored by terms describing pain severity extremes
Anterior flexion of shoulder joint (0-180°) | 0,1,2,4,8,12 weeks
  Passive activity of the shoulder joint
shoulder joint abduction (0-180°) | 0,1,2,4,8,12 weeks
  Passive activity of the shoulder joint
shoulder internal rotator (1-18 score) | 0,1,2,4,8,12 weeks
  The thumb tip reaches the highest point of the back cone:Score1-12: T1-T12; Score13-17:L1-L5;18: below the sacrum;
shoulder external rotator (0-180°) | 0,1,2,4,8,12 weeks
  Passive activity of the shoulder joint

CONTACTS AND LOCATIONS:
Overall Officials: Pintong Huang, Principal Investigator — Department of Ultrasound in Medicine, The Second Affiliated AHospital of Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
I'd like to share the IPD with the other researchers after the paper is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: I'd like to share the IPD with the other researchers after the paper is published.

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT04931511/SAP_000.pdf